CLINICAL TRIAL: NCT07179042
Title: A Pilot Study to Assess the Feasibility of a Randomized, Double-blind, Placebo-controlled Trial Investigating Intertrochanteric Femur Fracture Patients Who Receive Metformin With a Placebo
Brief Title: Intertrochanteric Femur Fracture Patients Who Receive Metformin With a Placebo
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 189701
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Intertrochanteric Femur Fracture; Muscle Atrophy
Keywords: Intertrochanteric Femur Fracture; Muscle Atrophy; Metformin; Randomized; Double-blind; Placebo-controlled trial
MeSH Terms: conditions — Muscular Atrophy | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Randomized, double-blind, placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo tablets (Placebo Comparator): Encapsulated placebo tablets per day (dosage for days 1-7 following the surgery is 500 mg/day, days 8-13 is 1000 mg/day, days 14-119 is 1500 mg/day).
  Interventions: Drug: Placebo
- Metformin tablets (Experimental): Encapsulated Metformin tablets per day (dosage for days 1-7 following the surgery is 500 mg/day, days 8-13 is 1000 mg/day, days 14-119 is 1500 mg/day).
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo — Placebo tablets will be dispensed to the participants for 119-days.
  Arms: Placebo tablets
Drug: Metformin — Metformin tablets will be dispensed to the participants for 119-days.
  Other Names: Glucophage, Glumetza, Riomet, Fortamet, and N,N-dimethylbiguanide
  Arms: Metformin tablets

SUMMARY:
The investigators central hypothesis is that metformin supplementation will be well-tolerated, safe, and provide patients with improved functional and muscle morphology outcomes following intertrochanteric femur fracture. The objectives will be tested in older adults that sustain a hip fracture and are randomized to receive a daily oral dose (1.5g daily) of metformin or a non-active placebo during 4 months of recovery following surgery.

DETAILED DESCRIPTION:
This study team investigates a patient population that undergoes muscle atrophy and falls under the current IND indication of metformin usage to prevent muscle atrophy and enhance muscle growth. The investigators are now proposing to utilize metformin as a novel tool to enhance muscle recovery following a hip fracture in older adults. The investigators currently preparing an IRB protocol in which we plan to perform a pilot study where older adult hip fracture patients are randomized to metformin or placebo. The investigators propose to use metformin to help enhance muscle recovery outcomes in this experimental study design since there are no effective methods to maximize muscle regrowth in older adults following hip fracture.

Hip fracture is a common and costly injury for hundreds of thousands of U.S. older adults every year resulting in devastating health consequences for many. Muscle atrophy is evident at 1 month post-surgery and commonly persists at least 2-6 months afterwards. This is alarming considering that many are considered sarcopenic leaving little muscle reserve to spare to maintain physical function in this population. Consequently, many are not likely to return to pre-fracture functional level one year after fracture. Rehabilitation strategies following hip fracture has remained largely unchanged over the past several decades, suggesting that older adults recovering from hip fracture could benefit from new, innovative approaches that target muscle mass and function.

Local inflammation has received considerable attention as an underlying mechanism contributing to a decline in skeletal muscle health of older adults with physical function deficits. Skeletal muscle inflammation is heightened in older adults and further in older adults who are inactive. Therefore, it is not surprising that the severe physical trauma and associated physical inactivity that accompanies recovery from hip fracture surgery is characterized by a robust muscle inflammatory response as numerous investigators have previously noted. Though inflammation is clearly important for proper muscle regeneration, hyper- and prolonged inflammation can lead to atrophy possibly interfering with muscle and functional recovery in older adults after hip fracture. Indeed, senescent cells, defined as a state of cell-cycle arrest, are a source of inflammation and accumulate in muscle tissue during injury thereby impairing tissue function. Aging further heightens the accumulation of senescent cells due to poor removal by immune cells given that the immune system declines with age.

Metformin has gained attention for exerting pleiotropic effects targeting key hallmarks of aging. However, the role of metformin on regulating muscle cell size and function in patients following hip fracture is unknown. Metformin has recently been shown to lessen cellular senescence burden in a variety of cell and tissue types in experimental cell culture and rodent models. Metformin may preserve muscle mass by activating AMPKα thereby limiting skeletal muscle inflammation through pro-inflammatory pathways such as NFκB and TLR4 signaling. In prior rodent studies, metformin has shown to attenuate muscle atrophy, muscle proteolysis, and fibrosis during muscle wasting conditions. Moreover, metformin has been shown to increase satellite cell proliferation and improve muscle regeneration following burn injury in mice and reduce muscle fibrosis induced by knee joint immobilization in rat. Importantly, we have recently shown that a clinical dose of metformin given to older adults on bed rest was a safe and effective strategy to improve muscle recovery by reducing tissue fibrosis and muscle inflammation and senescent cell accumulation suggesting that such an approach may likewise show promising outcomes in patients recovering from hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 60y and older.
* Displaced hip fracture (femoral neck, intertrochanteric femur, subtrochanteric femur fracture).
* Low energy mechanism of injury (ground level fall, etc).
* Operative treatment within 72 hours of injury.
* Previously ambulatory.

Exclusion Criteria:

* History of kidney disease or failure (CKD > stage 4; eGFR < 45 mL/min/1.73m2).
* History of diabetes mellitus (HbA1c > 6.5).
* Associated lower extremity fracture (ipsilateral or contralateral).
* Pathologic fracture.
* Presence of infection at the fracture site.
* History of metabolic bone disease (Pagets, etc.).
* Severe cognitive impairment (Six Item Screener with 3 or more errors).
* Stage 5 Parkinson's Disease.
* Open fracture.
* Risk of developing metformin-associated hypoglycemia (e.g., hepatic impairment (by history or screening laboratory assessment), presence of hypoglycemia at screening, history of adrenal or pituitary insufficiency, alcohol use disorder, subjects unable to maintain normal oral intake).
* Severe hepatic impairment (Child-Pugh C).
* Expected survival < 6 months (based on clinical judgement).

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Mid-thigh size (MTS), (centimeters) | 2-weeks after surgery
  Mid-thigh circumference will be assessed in the participants. These tests will occur during the standard clinical follow-up visits at 2, 8, and 16 weeks. Each participant will have both legs assessed.
Mid-thigh size (MTS), (centimeters) | 8-weeks after surgery
  Mid-thigh circumference will be assessed in the participants. These tests will occur during the standard clinical follow-up visits at 2, 8, and 16 weeks. Each participant will have both legs assessed.
Mid-thigh size (MTS), (centimeters) | 16-weeks after surgery
  Mid-thigh circumference will be assessed in the participants. These tests will occur during the standard clinical follow-up visits at 2, 8, and 16 weeks. Each participant will have both legs assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States